Official Title of Study: Alcohol PBS and Thinking about the Past

**NCT Number:** Not Assigned

Unique Protocol ID: IRB20201070D

**Date of Document:** 09/10/2021

## **Planned Analysis**

Statistical Design: The statistical design uses a multilevel structural equation model. The model will compare three conditions: Negative Event, Negative Event w/ a detailed description of the event, Negative Event w/ generated Counterfactuals to reduce future negative events, and Protective Behavioral Strategy Personalized Normative Feedback (PBS-PNF). Each condition will be used to predict protective behavioral strategies. Protective behavioral strategies will then predict alcohol and alcohol consequences. As the conditions are at the between-subject level, the hypotheses are specific to between subject effects, however, the data will be modeled at both the within- and between- subjects level (see Figure 1). In order to decompose variance across levels, all level 1 variables will be centered at the person level while all level 2 variables will be centered at the grandmean. Only weeks during which participants consume alcohol will be included in the analysis, as the intervention target (PBS) only occurs on drinking days.

<u>Covariates:</u> At level 1, we will control for week of study and number of drinking days. At level 2 we will control for biological sex at birth.

**Hypothesis 1:** Relative to control, the counterfactual condition will result in significantly more use of PBS during drinking days and will be *at least* non-inferior to PBS personalized normative feedback (significant effect of path a).

**Hypothesis 2:** Relative to control, the counterfactual condition will exert a significant specific indirect effect on alcohol problems through PBS (H2 = path a x path b).

**Hypothesis 3:** Relative to control, the counterfactual condition will exert a significant total indirect effect on alcohol problems through PBS use and alcohol use (H3 = H2 + [path a x path c x path d]).



## Mplus Code:

H3 = H2+(c\*d);

usevar are CFcondition PBSPNFcondition NegEventcondition L1PBS L1Drinks L2PBS L2Drinks Problems;

within are L1PBS L1Drinks: between are CFcondition PBSPNFcondition NegEventcondition L2PBS L2Drinks; cluster = ID; analysis: estimator = mlr; PROCESSORS = 2: type = twolevel; model: %within% L1Drinks on L1PBS; Problems on L1Drinks L1PBS: [L1Drinks @0]; [L1PBS @0]; %between% L2PBS on CFcondition(a); L2PBS on PBSPNFcondition: L2PBS on NegEventcondition; L2Drinks on L2PBS(c); Problems on L2PBS(b); Problems on L2Drinks(d); Model Constraint: New(H1 H2 H3); H1 = a: H2 = a\*b

**Exploratory Analysis:** We will examine differences between the counterfactual condition and PBS PNF condition to determine equivalence between the two intervention effects. This approach will use a two one-sided equivalence test (TOST), to compare the two active treatments (Lakens, 2017). This allows for a comparison of a new treatment against the observed effects of an existing treatment (rather than against the traditional null hypothesis). In doing so, we will specify an "equivalence" margin of Cohen's *d* -0.20 to 0.20 (a small effect in both directions). We will then calculate 95% confidence intervals of the effect size difference between the Counterfactual and PBS-PNF. A positive value indicates a stronger effect of Counterfactual relative to PBS PNF, while a negative value indicates a weaker effect. This approach allows for the statistical determination of whether the observed effect is equivalent to the standard treatment, superior to the standard treatment.